CLINICAL TRIAL: NCT00752232
Title: A Phaseiia, Multicenter, Randomized, Third-party Unblinded, Adjuvant And Placebo-controlled, Multiple Ascending Dose, Safety, Tolerability And Immunogenicity Trial Of Acc-001 And Qs-21 Adjuvant In Japanese Subjects With Mild To Moderate Alzheimer's Disease.
Brief Title: Study Evaluating ACC-001 in Japanese Patients With Mild To Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: JANSSEN Alzheimer Immunotherapy Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3134K1-2202; B2571006 (Other: Alias Study Number)
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Results first posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-11

CONDITIONS: Alzheimer Disease
Keywords: Phase IIa; multiple ascending dose study of ACC-001
MeSH Terms: conditions — Alzheimer Disease | interventions — vanutide cridificar; saponin QA-21V1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ACC-001+QS-21 (Experimental): Active vaccine + adjuvant, IM injection, dose of 3, 10, 30 micrograms, Day 1, month 3, 6, 9, 12
  Interventions: Biological: ACC-001; Other: QS-21
- ACC-001 (Experimental): Active vaccine, IM injection, dose of 3, 10, 30 micrograms, Day 1, month 3, 6, 9, 12
  Interventions: Biological: ACC-001
- QS-21 (Placebo Comparator): Adjuvant, IM injection, dose of 50 micrograms, Day 1, month 3, 6, 9, 12
  Interventions: Other: QS-21
- PBS (Placebo Comparator): Placebo, IM injection, Day 1, month 3, 6, 9, 12
  Interventions: Other: PBS

INTERVENTIONS:
Biological: ACC-001 — IM injection, dose of 3, 10, 30 micrograms, Day 1, month 3, 6, 9, 12
  Arms: ACC-001+QS-21
Other: QS-21 — IM injection, dose of 50 micrograms, Day 1, month 3, 6, 9, 12
  Arms: ACC-001+QS-21
Biological: ACC-001 — IM injection, dose of 3, 10, 30 micrograms, Day 1, month 3, 6, 9, 12
  Arms: ACC-001
Other: QS-21 — IM injection, dose of 50 micrograms, Day 1, month 3, 6, 9, 12
  Arms: QS-21
Other: PBS — IM injection, Day 1, month 3, 6, 9, 12
  Arms: PBS

SUMMARY:
The study is to evaluate the safety, tolerability and whether there is an immune system response to multiple doses of ACC-001 with or without the use of a substance that may increase the response to the drug.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild to moderate Alzheimer's Disease
* Mini Mental Status Exam (MMSE) of 16-26

Exclusion Criteria:

* Significant Neurological Disease
* Major Psychiatric Disorder
* Clinically significant systemic illness

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- Japan (10):
  - Suwa Red Cross Hospital, Suwa, Nagano
  - Tazuke Kofukai Medical Research Institute Kitano Hospital, Osaka, Osaka
  - Osaka Medical College Hospital, Takatsuki, Osaka
  - Meitetsu Hospital, Aichi
  - Ibaraki Prefectural Central Hospital, Ibaraki
  - Shonan Atsugi Hospital, Kanagawa
  - Kitasato University East Hospital, Kanagawa
  - Juntendo University Hospital, Tokyo
  - Juntendo Tokyo Koto Geriatric Medical Center, Tokyo
  - Kanto Ctrl Hp of the Mutual Aid Asso of Public school Teache, Tokyo

REFERENCES:
- [Derived] Arai H, Suzuki H, Yoshiyama T. Vanutide cridificar and the QS-21 adjuvant in Japanese subjects with mild to moderate Alzheimer's disease: results from two phase 2 studies. Curr Alzheimer Res. 2015;12(3):242-54. doi: 10.2174/1567205012666150302154121. PMID 25731629
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3134K1-2202&StudyName=Study%20Evaluating%20ACC-001%20in%20Japanese%20Patients%20With%20Mild%20To%20Moderate%20Alzheimer%27s%20Disease

RESULTS

PARTICIPANT FLOW:
Groups:
- ACC-001 3 Micrograms +QS-21: A cohort of participants who received intramuscular (IM) injection of active vaccine ACC-001 (3 micrograms) + adjuvant QS-21 (50 micrograms) at Day 1, month 3, 6, 9 and 12
- ACC-001 10 Micrograms: A cohort of participants who received IM injection of active vaccine ACC-001 (10 micrograms) at Day1, month 3, 6, 9 and 12
- ACC-001 10 Micrograms + QS-21: A cohort of participants who received IM injection of active vaccine ACC-001 (10 micrograms) + adjuvant QS-21 (50 micrograms) at Day
  1, month 3, 6, 9 and 12
- ACC-001 30 Micrograms: A cohort of participants who received IM injection of active vaccine ACC-001 (30 micrograms) at Day 1, month 1, 3, 6 and 12
- ACC-001 30 Micrograms +QS-21: A cohort of participants who received IM injection of active vaccine ACC-001 (30 micrograms) + adjuvant QS-21 (50 micrograms) at Day 1, month 1, 3, 6 and 12
- QS-21: A cohort of participants who received IM injection of adjuvant QS-21 (50 micrograms) at Day 1, month 3, 6, 9 and 12
- Phosphate Buffered Saline (PBS): A cohort of participants who received phosphate buffered saline (PBS) at Day 1, month 3, 6, 9 and 12
Period: Overall Study
Arm/Group | ACC-001 3 Micrograms +QS-21 | ACC-001 10 Micrograms | ACC-001 10 Micrograms + QS-21 | ACC-001 30 Micrograms | ACC-001 30 Micrograms +QS-21 | QS-21 | Phosphate Buffered Saline (PBS)
Started | 6 | 6 | 6 | 6 | 6 | 6 | 4
Completed | 4 | 6 | 5 | 5 | 3 | 5 | 4
Not Completed | 2 | 0 | 1 | 1 | 3 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Caregiver request | 2 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Investigator request | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Subject request | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Group home admission | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Caregiver could not attend the subject | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACC-001 3 Micrograms +QS-21 | ACC-001 10 Micrograms | ACC-001 10 Micrograms + QS-21 | ACC-001 30 Micrograms | ACC-001 30 Micrograms +QS-21 | QS-21 | Phosphate Buffered Saline (PBS) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 4 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.33 (9.35) | 69.50 (6.92) | 73.00 (7.67) | 70.17 (3.13) | 66.00 (10.79) | 67.00 (9.19) | 69.50 (4.80) | 69.50 (7.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5 | 4 | 2 | 4 | 3 | 23
  Male | 5 | 2 | 1 | 2 | 4 | 2 | 1 | 17

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-emergent Adverse Events (AEs) by Severity
Description: Number of participants who experienced mild, moderate, or severe AEs (mild = does not interfere with subject's usual function; moderate = interferes to some extent with subject's usual function; severe = interferes significantly with subject's usual function)
Time Frame: Baseline up to 24 months
Population: The safety analysis population includes all of the randomly assigned participants who took at least one dose of study medication.
Measure: Number; unit: Participants
Groups:
- ACC-001 10 Micrograms + QS-21: A cohort of participants who received IM injection of active vaccine ACC-001 (10 micrograms) + adjuvant QS-21 (50 micrograms) at Day1, month 3, 6, 9 and 12
Arm/Group | ACC-001 3 Micrograms +QS-21 | ACC-001 10 Micrograms | ACC-001 10 Micrograms + QS-21 | ACC-001 30 Micrograms | ACC-001 30 Micrograms +QS-21 | QS-21 | Phosphate Buffered Saline (PBS)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 4
Participants
  Mild | 5 | 6 | 4 | 5 | 3 | 6 | 3
  Moderate | 0 | 0 | 0 | 1 | 2 | 0 | 0
  Severe | 1 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Brain Abnormalities in Magnetic Resonance Imaging (MRI) Data
Description: Number of participants with brain abnormalities in MRI data that are either consistent or not consistent with AD, as determined by investigator.
Time Frame: Baseline up to 24 months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | ACC-001 3 Micrograms +QS-21 | ACC-001 10 Micrograms | ACC-001 10 Micrograms + QS-21 | ACC-001 30 Micrograms | ACC-001 30 Micrograms +QS-21 | QS-21 | Phosphate Buffered Saline (PBS)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 4
Participants
  Abnormal-inconsistent with AD | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Abnormal-consistent with AD | 6 | 6 | 6 | 6 | 6 | 5 | 4

3. Primary Outcome: Number of Participants With Abnormalities in Neurological Examination
Description: Number of participants with abnormalities in neurological examinations as determined by the investigators. Neurological examinations included Mental Status, Speech, Cranial Nerves (including pupil equality and reactivity), Visual field, Sensory, Motor, Coordination, Gait, Primitive reflexes, Tendon reflexes and Romberg.
Time Frame: Baseline up to 24 months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | ACC-001 3 Micrograms +QS-21 | ACC-001 10 Micrograms | ACC-001 10 Micrograms + QS-21 | ACC-001 30 Micrograms | ACC-001 30 Micrograms +QS-21 | QS-21 | Phosphate Buffered Saline (PBS)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 4
Participants
  Total | 2 | 0 | 1 | 0 | 0 | 0 | 0
  Mental Status | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Speech | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Cranial Nerves | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Visual field | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sensory | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Motor | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Coordination | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Gait | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Primitive reflexes | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Tendon reflexes | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Romberg | 0 | 0 | 1 | 0 | 0 | 0 | 0

4. Secondary Outcome: Anti-a-beta IgG Titer at Specified Visits
Description: Geometric mean of anti-a-beta IgG titer from pre-study through Week 104
Time Frame: Baseline up to 24 months
Population: The population for immunogenicity analysis includes all of the randomly assigned participants who took at least one dose of study medication, having the baseline and at least one post baseline immunogenicity evaluation.
Measure: Geometric Mean (95% Confidence Interval); unit: Units/mL
Arm/Group | ACC-001 3 Micrograms +QS-21 | ACC-001 10 Micrograms | ACC-001 10 Micrograms + QS-21 | ACC-001 30 Micrograms | ACC-001 30 Micrograms +QS-21 | QS-21 | Phosphate Buffered Saline (PBS)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 4
Units/mL
  Pre-study (n=6, 6, 6, 6, 6, 6, 4) | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 2 (n=6, 6, 6, 6, 6, 6, 4) | 62.3 [35.4 to 110.0] | 50.0 [50.0 to 50.0] | 86.1 [21.3 to 347.9] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 6 (n=6, 6, 6, 6, 6, 6, 4) | 65.3 [32.9 to 129.7] | 50.0 [50.0 to 50.0] | 105.4 [43.4 to 255.8] | 50.0 [50.0 to 50.0] | 58.9 [38.7 to 89.5] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 10 (n=6, 6, 5, 6, 6, 6, 4) | 70.9 [28.9 to 174.4] | 50.0 [50.0 to 50.0] | 93.5 [28.8 to 303.0] | 59.2 [38.3 to 91.5] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 14 (n=6, 6, 5, 6, 6, 5, 4) | 2468.3 [775.0 to 7861.2] | 50.0 [50.0 to 50.0] | 8976.5 [680.6 to 118398.0] | 163.7 [29.5 to 908.5] | 2166.0 [390.7 to 12007.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 16 (n=6, 6, 5, 6, 6, 5, 4) | 1383.1 [340.9 to 5612.4] | 50.0 [50.0 to 50.0] | 4886.1 [348.5 to 68510.7] | 135.9 [25.6 to 720.8] | 1506.4 [297.6 to 7623.9] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 24 (n=6, 6, 5, 6, 6, 5, 4) | 476.2 [54.7 to 4148.3] | 50.0 [50.0 to 50.0] | 1427.3 [80.1 to 25425.0] | 113.4 [29.4 to 436.7] | 518.9 [91.4 to 2938.6] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 28 (n=6, 6, 5, 6, 6, 5, 4) | 3025.4 [1089.9 to 8398.6] | 50.0 [50.0 to 50.0] | 6815.7 [180.5 to 257414.9] | 324.6 [28.3 to 3728.9] | 7088.0 [1939.0 to 25910.8] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 30 (n=6, 6, 5, 6, 6, 5, 4) | 2340.1 [715.0 to 7659.1] | 50.0 [50.0 to 50.0] | 6016.6 [190.4 to 190127.4] | 287.6 [24.6 to 3359.6] | 5989.4 [1366.6 to 26250.5] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 34 (n=6, 6, 5, 6, 6, 5, 4) | 1689.7 [371.7 to 7681.8] | 50.0 [50.0 to 50.0] | 5482.8 [194.8 to 154346.1] | 214.7 [26.1 to 1765.7] | 3730.2 [885.6 to 15711.5] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 38 (n=6, 6, 5, 6, 6, 5, 4) | 4806.1 [2395.8 to 9641.1] | 50.0 [50.0 to 50.0] | 5751.3 [301.4 to 109732.2] | 353.5 [33.0 to 3785.7] | 10540.9 [3111.3 to 35711.8] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 40 (n=6, 6, 5, 6, 6, 5, 4) | 5147.1 [2523.9 to 10496.7] | 50.0 [50.0 to 50.0] | 4215.3 [174.2 to 101984.8] | 288.1 [32.2 to 2573.6] | 8889.6 [2565.3 to 30805.1] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 50 (n=6, 6, 5, 6, 6, 5, 4) | 2083.4 [1077.9 to 4026.8] | 50.0 [50.0 to 50.0] | 2792.0 [144.6 to 53925.7] | 162.0 [31.3 to 839.0] | 4184.8 [921.0 to 19015.0] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 54 (n=4, 6, 5, 6, 6, 5, 4) | 7028.9 [1100.8 to 44879.8] | 50.0 [50.0 to 50.0] | 4316.0 [312.0 to 59700.9] | 467.9 [81.4 to 2689.7] | 12638.9 [5577.9 to 28638.3] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 56 (n=4, 6, 5, 6, 6, 5, 4) | 7274.7 [1037.3 to 51016.9] | 50.0 [50.0 to 50.0] | 3642.5 [175.7 to 75527.4] | 372.7 [78.5 to 1769.7] | 8644.2 [3365.0 to 22205.8] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 66 (n=5, 6, 5, 6, 6, 5, 4) | 3841.6 [825.2 to 17883.9] | 50.0 [50.0 to 50.0] | 3069.8 [165.5 to 56949.5] | 207.0 [46.8 to 915.6] | 4555.6 [1016.8 to 20411.1] | 147.9 [7.3 to 3006.4] | 50.0 [50.0 to 50.0]
  Week 78 (n=4, 6, 5, 5, 6, 5, 4) | 2599.1 [215.5 to 31342.0] | 50.0 [50.0 to 50.0] | 2236.1 [155.3 to 32198.4] | 231.0 [34.2 to 1559.2] | 2484.6 [571.3 to 10806.5] | 50.0 [50.0 to 50.0] | 50.0 [50.0 to 50.0]
  Week 91 (n=4, 0, 1, 0, 0, 1, 0) | 1870.6 [159.8 to 21900.7] | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | 2959.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | 50.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week.
  Week 104 (n=4, 0, 1, 0, 0, 1, 0) | 1403.1 [112.1 to 17561.2] | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | 2557.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | 50.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week.

5. Secondary Outcome: Anti-a-beta IgM Titer at Specified Visits
Description: Geometric mean of anti-a-beta IgM titer from pre-study through Week 104
Time Frame: Baseline up to 24 months
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Units/mL
Arm/Group | ACC-001 3 Micrograms +QS-21 | ACC-001 10 Micrograms | ACC-001 10 Micrograms + QS-21 | ACC-001 30 Micrograms | ACC-001 30 Micrograms +QS-21 | QS-21 | Phosphate Buffered Saline (PBS)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 4
Units/mL
  Pre-study (n=6, 6, 6, 6, 6, 6, 4) | 25.0 [25.0 to 25.0] | 31.7 [17.3 to 58.1] | 25.0 [25.0 to 25.0] | 32.9 [16.3 to 66.4] | 31.0 [17.8 to 53.9] | 36.1 [14.0 to 93.2] | 37.6 [10.3 to 137.9]
  Week 2 (n=6, 6, 6, 6, 6, 6, 4) | 38.0 [17.5 to 82.6] | 32.5 [16.5 to 63.9] | 56.6 [13.9 to 231.4] | 32.1 [16.9 to 60.7] | 116.6 [26.6 to 511.8] | 40.9 [16.2 to 103.2] | 38.0 [10.0 to 144.7]
  Week 6 (n=6, 6, 6, 6, 6, 6, 4) | 51.0 [15.9 to 163.5] | 34.9 [19.5 to 62.5] | 51.1 [15.8 to 165.2] | 37.9 [18.7 to 77.0] | 123.0 [25.9 to 584.8] | 41.2 [16.2 to 105.1] | 37.3 [10.4 to 133.4]
  Week 10 (n=6, 6, 5, 6, 6, 6, 4) | 53.7 [15.4 to 188.0] | 35.4 [19.5 to 64.4] | 58.6 [13.7 to 251.3] | 32.1 [16.9 to 61.0] | 128.4 [30.2 to 546.2] | 40.5 [17.3 to 94.9] | 37.4 [10.4 to 134.5]
  Week 14 (n=6, 6, 5, 6, 6, 5, 4) | 395.6 [12.8 to 12238.1] | 38.3 [18.9 to 77.5] | 357.1 [43.7 to 2920.6] | 52.6 [20.7 to 133.5] | 614.7 [125.8 to 3002.9] | 47.7 [14.9 to 153.3] | 97.1 [1.3 to 7277.6]
  Week 16 (n=6, 6, 5, 6, 6, 5, 4) | 380.4 [9.4 to 15415.0] | 37.6 [19.3 to 73.2] | 330.1 [48.0 to 2271.7] | 57.7 [20.7 to 161.0] | 683.8 [80.2 to 5829.6] | 46.3 [14.1 to 152.5] | 35.4 [11.7 to 107.6]
  Week 24 (n=6, 6, 5, 6, 6, 5, 4) | 204.0 [4.4 to 9434.1] | 34.7 [20.4 to 59.2] | 208.6 [44.6 to 975.7] | 58.8 [19.2 to 180.1] | 586.9 [60.2 to 5724.2] | 37.1 [12.4 to 110.6] | 35.9 [11.4 to 113.2]
  Week 28 (n=6, 6, 5, 6, 6, 5, 4) | 651.0 [47.9 to 8850.3] | 41.4 [17.7 to 96.6] | 356.7 [50.9 to 2501.4] | 77.7 [16.7 to 362.3] | 2706.8 [366.9 to 19970.2] | 58.6 [17.2 to 199.2] | 37.9 [10.1 to 142.4]
  Week 30 (n=6, 6, 5, 6, 6, 5, 4) | 949.1 [88.1 to 10223.9] | 40.6 [18.4 to 89.5] | 719.1 [81.7 to 6327.1] | 79.0 [17.9 to 349.3] | 3456.7 [381.6 to 31311.7] | 47.4 [22.9 to 98.0] | 39.4 [9.2 to 168.5]
  Week 34 (n=6, 6, 5, 6, 6, 5, 4) | 446.7 [20.4 to 9760.9] | 38.7 [19.0 to 78.6] | 666.0 [80.9 to 5481.4] | 62.3 [20.1 to 192.9] | 2182.0 [235.7 to 20199.3] | 43.2 [17.0 to 109.3] | 38.0 [10.0 to 144.7]
  Week 38 (n=6, 6, 5, 6, 6, 5, 4) | 473.5 [32.9 to 6813.1] | 39.1 [18.9 to 80.8] | 702.1 [201.8 to 2443.2] | 99.2 [24.6 to 400.2] | 2639.4 [368.5 to 18904.8] | 48.8 [22.1 to 107.8] | 39.4 [9.3 to 167.3]
  Week 40 (n=6, 6, 5, 6, 6, 5, 4) | 509.6 [38.5 to 6736.7] | 38.0 [19.2 to 75.2] | 574.8 [192.7 to 1714.8] | 83.6 [19.0 to 367.4] | 2545.5 [313.6 to 20661.2] | 45.9 [21.8 to 96.6] | 37.0 [10.6 to 128.9]
  Week 50 (n=6, 6, 5, 6, 6, 5, 4) | 223.8 [15.2 to 3301.7] | 37.8 [18.8 to 76.1] | 432.4 [140.8 to 1328.1] | 71.5 [27.0 to 189.3] | 1418.2 [230.1 to 8741.4] | 61.2 [29.1 to 128.6] | 38.2 [9.9 to 146.9]
  Week 54 (n=4, 6, 5, 6, 6, 5, 4) | 836.2 [4.7 to 147881.4] | 37.9 [19.2 to 74.8] | 450.0 [186.4 to 1086.3] | 140.9 [25.3 to 782.7] | 1668.1 [309.0 to 9005.8] | 51.2 [21.4 to 122.5] | 36.5 [10.9 to 122.2]
  Week 56 (n=4, 6, 5, 6, 6, 5, 4) | 678.8 [4.3 to 108248.9] | 36.9 [19.6 to 69.6] | 422.3 [180.7 to 986.6] | 119.4 [18.3 to 780.5] | 1507.7 [309.5 to 7344.5] | 42.4 [17.0 to 105.3] | 34.6 [12.3 to 97.6]
  Week 66 (n=5, 6, 5, 6, 6, 5, 4) | 371.0 [16.3 to 8454.7] | 37.1 [19.4 to 71.0] | 331.1 [131.3 to 834.6] | 105.3 [15.9 to 698.4] | 1058.7 [226.9 to 4939.1] | 56.3 [12.7 to 249.0] | 35.4 [11.7 to 106.5]
  Week 78 (n=4, 6, 5, 5, 6, 5, 4) | 450.1 [6.9 to 29432.6] | 39.9 [18.6 to 85.5] | 209.8 [81.9 to 537.8] | 134.2 [13.3 to 1357.2] | 759.3 [135.9 to 4242.2] | 32.7 [15.6 to 68.5] | 34.1 [12.7 to 92.1]
  Week 91 (n=4, 0, 1, 0, 0, 1, 0) | 321.8 [5.8 to 17755.5] | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | 60.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | 25.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week.
  Week 104 (n=4, 0, 1, 0, 0, 1, 0) | 226.1 [4.6 to 11037.7] | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | 54.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week. | 25.0 [NA to NA] — 95% confidence interval was not estimable since only one participant was evaluable. | NA [NA to NA] — Data were not analyzed as no participants were evaluable for the particular week.

6. Other Pre Specified Outcome: The Mean Changes in Alzheimer's Disease Assessment Scale-Cognitive Behavior (ADAS-Cog) Score From Baseline at Week 12, 26, 36, 52, 78 and 104.
Description: The ADAS-Cog is a 12-item,objective measure of cognitive function, consisting of 1) Word Recall, 2) Naming Objects and Fingers, 3) Following Commands, 4) Constructional Praxis, 5) Ideational Praxis, 6) Orientation, 7) Word Recognition, 8) Recall of Test Instructions, 9) Spoken Language Ability, 10) Word-Finding Difficulty, 11) Comprehension of Spoken Language and 12) Concentration/Distractibility. For this stuy, the ADAS-Cog total score is derived by summing the individual scores from items 1 to 11. Total score ranges from 0 to 70 points, with higher scores indicating a greater degree of impairment.
Time Frame: Baseline up to 24 months
Population: Efficacy analyses were performed on the modified intent-to-treat (mITT) population. The mITT population included all of the randomly assigned participants who took at least one dose of study medication, and had the baseline and at least one post baseline evaluation of the key efficacy variable (ADAS-Cog).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | ACC-001 3 Micrograms +QS-21 | ACC-001 10 Micrograms | ACC-001 10 Micrograms + QS-21 | ACC-001 30 Micrograms | ACC-001 30 Micrograms +QS-21 | QS-21 | Phosphate Buffered Saline (PBS)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 4
Units on a scale
  Week 12 (n=6, 6, 5, 6, 6, 6, 4) | 4.06 (6.45) | -2.00 (2.86) | 1.93 (5.51) | -0.94 (2.72) | -1.28 (3.74) | 1.28 (4.95) | 2.92 (1.13)
  Week 26 (n=6, 6, 5, 6, 6, 5, 4) | 2.22 (4.88) | 0.78 (4.63) | -1.20 (1.17) | 1.67 (4.30) | -1.78 (2.45) | 1.93 (9.59) | 1.33 (3.27)
  Week 36 (n=6, 6, 5, 6, 6, 5, 4) | 4.89 (7.53) | -0.50 (2.75) | -0.93 (1.53) | 0.56 (3.94) | -1.17 (4.88) | 2.93 (5.08) | 3.92 (4.15)
  Week 52 (n=6, 6, 5, 6, 6, 5, 4) | 5.83 (9.41) | -2.56 (4.18) | -1.73 (2.24) | 3.56 (4.81) | -2.00 (3.75) | 5.80 (7.39) | 0.92 (2.60)
  Week 78 (n=4, 6, 5, 5, 6, 5, 4) | 8.50 (10.09) | -0.33 (3.03) | -0.07 (4.23) | 2.47 (3.90) | -0.06 (5.16) | 6.47 (12.32) | 4.50 (4.39)
  Week 104 (n=4, 0 1, 0, 0, 1, 0) | 5.92 (8.86) | NA (NA) — Data were not analyzed as no participants were evaluable for the particular week. | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data were not analyzed as no participants were evaluable for the particular week. | NA (NA) — Data were not analyzed as no participants were evaluable for the particular week. | 6.33 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data were not analyzed as no participants were evaluable for the particular week.

7. Other Pre Specified Outcome: The Mean Changes in Disability Assessment for Dementia (DAD) Score From Baseline at Week 12, 26, 36, 52, 78 and 104.
Description: The DAD is administered through an interview with the caregiver and measures instrumental and basic activities of daily living. A total score is obtained by adding the rating for each question and converting this total score out of 100. Higher scores represent less disability in ADL while lower scores indicate more dysfunction.
Time Frame: Baseline up to 24 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | ACC-001 3 Micrograms +QS-21 | ACC-001 10 Micrograms | ACC-001 10 Micrograms + QS-21 | ACC-001 30 Micrograms | ACC-001 30 Micrograms +QS-21 | QS-21 | Phosphate Buffered Saline (PBS)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 4
Units on a scale
  Week 12 (n=4, 5, 4, 6, 5, 5, 4) | 0.8 (4.1) | -0.8 (3.6) | 5.1 (7.4) | -3.5 (7.0) | -3.0 (11.8) | -8.8 (10.8) | 3.9 (6.8)
  Week 26 (n=4, 4, 4, 6, 5, 5, 4) | 2.1 (9.5) | 1.8 (5.3) | 6.8 (6.8) | -1.8 (6.9) | -0.6 (3.3) | -5.4 (13.2) | 4.1 (16.0)
  Week 36 (n=4, 4, 5, 6, 5, 5, 4) | 1.4 (9.1) | 4.9 (6.9) | 3.7 (4.4) | -2.7 (6.3) | -1.7 (9.3) | -6.8 (11.5) | -1.4 (15.1)
  Week 52 (n=4, 5, 5, 6, 5, 5, 4) | -7.8 (15.6) | -3.3 (21.7) | 4.2 (5.3) | -8.3 (21.0) | 0.8 (16.1) | -11.4 (9.1) | 2.8 (10.4)
  Week 78 (n=2, 5, 4, 5, 5, 5, 4) | -12.0 (3.8) | -16.7 (26.5) | -1.3 (9.0) | -2.9 (9.7) | -1.0 (12.4) | -14.4 (10.0) | 3.4 (9.3)
  Week 104 (n=2, 0, 1, 0, 0, 1, 0) | -0.8 (1.2) | NA (NA) — Data were not analyzed as no participants were evaluable for the particular week. | 0.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data were not analyzed as no participants were evaluable for the particular week. | NA (NA) — Data were not analyzed as no participants were evaluable for the particular week. | -32.5 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data were not analyzed as no participants were evaluable for the particular week.

8. Other Pre Specified Outcome: The Mean Changes in Neuropsychological Test Battery (NTB) Score From Baseline at Week 12, 26, 36, 52, 78 and 104.
Description: The NTB is a composite of nine widely used neuropsychological tests that assess immediate and delayed recall of verbal and visual information, attention, verbal fluency and executive function. The cognitive tests included in the NTB are the Wechsler Memory Scale (WMS) Visual-Paired Associates (immediate and delayed), WMSVerbal Paired Associates (immediate and delayed), Rey Auditory Verbal Learning Test (immediate and delayed), WMS-Digit Span, Controlled Word Association Test, and Category Fluency Test. The NTB z-score is used for analysis. The z-score for each component is calculated through the following formula: z = (y_visit - y_base)/SD_base, where y_visit is a value at a particular time point and y_base is the average test score, and SD_base is the SD based on all participants' observed baseline scores in the study.
Time Frame: Baseline up to 24 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | ACC-001 3 Micrograms +QS-21 | ACC-001 10 Micrograms | ACC-001 10 Micrograms + QS-21 | ACC-001 30 Micrograms | ACC-001 30 Micrograms +QS-21 | QS-21 | Phosphate Buffered Saline (PBS)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 4
Z-score
  Week 12 (n=6, 6, 5, 6, 6, 6, 4) | 0.048 (0.314) | 0.002 (0.198) | 0.043 (0.306) | 0.030 (0.220) | -0.007 (0.266) | 0.058 (0.226) | 0.203 (0.092)
  Week 26 (n=6, 6, 5, 6, 6, 5, 4) | 0.114 (0.378) | -0.028 (0.420) | 0.272 (0.148) | 0.095 (0.404) | 0.374 (0.278) | 0.121 (0.180) | 0.215 (0.449)
  Week 36 (n=6, 6, 5, 6, 6, 5, 4) | 0.148 (0.573) | 0.188 (0.219) | 0.367 (0.222) | 0.267 (0.294) | 0.232 (0.388) | 0.061 (0.353) | 0.465 (0.494)
  Week 52 (n=6, 6, 5, 6, 6, 5, 4) | 0.171 (0.585) | 0.183 (0.274) | 0.247 (0.189) | -0.036 (0.312) | 0.255 (0.454) | 0.184 (0.320) | 0.411 (0.357)
  Week 78 (n=4, 6, 5, 5, 6, 5, 4) | 0.138 (0.597) | -0.047 (0.291) | 0.132 (0.261) | -0.160 (0.332) | 0.246 (0.515) | 0.184 (0.631) | 0.258 (0.399)
  Week 104 (n=4, 0, 1, 0, 0, 1, 0) | 0.048 (0.647) | NA (NA) — Data were not analyzed as no participants were evaluable for the particular week. | 0.345 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data were not analyzed as no participants were evaluable for the particular week. | NA (NA) — Data were not analyzed as no participants were evaluable for the particular week. | 0.118 (0.118) | NA (NA) — Data were not analyzed as no participants were evaluable for the particular week.

9. Other Pre Specified Outcome: The Mean Changes in Mini-Mental State Examination (MMSE) Score From Baseline at Week 4, 8, 12, 16, 26, 30, 36, 40, 52, 78 and 104.
Description: The MMSE is a brief, structured examination of cognitive function. It has a total score of 30 points (0-30), and any score equal to or lower than 26 points indicates cognitive impairment.
Time Frame: Baseline up to 24 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | ACC-001 3 Micrograms +QS-21 | ACC-001 10 Micrograms | ACC-001 10 Micrograms + QS-21 | ACC-001 30 Micrograms | ACC-001 30 Micrograms +QS-21 | QS-21 | Phosphate Buffered Saline (PBS)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 4
Units on a scale
  Week 4 (n=6, 6, 5, 6, 6, 6, 4) | -0.8 (2.6) | -0.2 (2.7) | 1.8 (2.5) | 1.0 (1.7) | 1.5 (2.4) | 1.0 (2.1) | 1.0 (2.4)
  Week 8 (n=6, 6, 5, 6, 6, 6, 4) | 0.5 (2.3) | 0.8 (2.8) | 1.4 (2.5) | 1.8 (1.6) | 2.0 (1.7) | 1.0 (2.7) | -0.3 (1.7)
  Week 12 (n=6, 6, 5, 6, 6, 6, 4) | -0.2 (3.6) | 0.3 (2.7) | -0.6 (2.5) | 0.8 (2.1) | 2.3 (2.9) | 0.7 (2.2) | 0.5 (2.4)
  Week 16 (n=6, 6, 5, 6, 6, 5, 4) | -0.2 (2.4) | 0.0 (1.1) | -0.6 (2.9) | 2.8 (1.6) | 1.2 (3.1) | 1.0 (4.3) | 0.3 (3.2)
  Week 26 (n=6, 6, 5, 6, 6, 5, 4) | -1.0 (4.7) | 0.5 (1.6) | 0.4 (3.6) | 0.3 (1.5) | 0.2 (2.9) | 0.2 (2.8) | 0.5 (3.1)
  Week 30 (n=6, 6, 5, 6, 6, 5, 4) | -1.3 (4.4) | 0.5 (1.8) | -1.6 (4.3) | 1.2 (1.3) | 1.3 (2.2) | 1.4 (4.1) | 0.3 (2.1)
  Week 36 (n=6, 6, 5, 6, 6, 5, 4) | -3.0 (5.8) | 0.0 (2.9) | 0.0 (2.3) | 0.8 (1.6) | 2.2 (2.8) | -0.2 (2.2) | -0.5 (3.1)
  Week 40 (n=6, 6, 5, 6, 6, 5, 4) | -2.5 (4.3) | 1.3 (4.2) | -0.4 (4.8) | 1.8 (1.7) | 1.8 (1.5) | 0.6 (2.1) | -2.3 (3.6)
  Week 52 (n=6, 6, 5, 6, 6, 5, 4) | -2.7 (5.4) | -0.3 (2.0) | -1.6 (3.4) | -0.3 (3.6) | 1.8 (2.6) | -0.8 (4.2) | -1.5 (1.7)
  Week 78 (n=4, 6, 5, 5, 6, 5, 4) | -4.8 (6.8) | -0.8 (4.5) | -1.2 (2.2) | -0.8 (1.9) | 0.3 (2.3) | -2.0 (2.9) | 0.3 (2.6)
  Week 104 (n=4, 0, 1, 0, 0, 1, 0) | -4.3 (7.4) | NA (NA) — Data were not analyzed as no participants were evaluable for the particular week. | 4.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data were not analyzed as no participants were evaluable for the particular week. | NA (NA) — Data were not analyzed as no participants were evaluable for the particular week. | -6.0 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data were not analyzed as no participants were evaluable for the particular week.

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- ACC-001 30 Micrograms: A cohort of participants who received IM injection of active vaccine ACC-001 (30 micrograms) at Day 1, month 3, 6, 9 and 12
- ACC-001 30 Micrograms + QS-21: A cohort of participants who received IM injection of active vaccine ACC-001 (30 micrograms) + adjuvant QS-21 (50 micrograms) at Day 1, month 1, 3, 6 and 12
Arm/Group | ACC-001 3 Micrograms +QS-21 | ACC-001 10 Micrograms | ACC-001 10 Micrograms + QS-21 | ACC-001 30 Micrograms | ACC-001 30 Micrograms + QS-21 | QS-21 | Phosphate Buffered Saline (PBS)
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 0/6 | 0/6 | 1/6 | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 4/6 | 6/6 | 5/6 | 6/6 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACC-001 3 Micrograms +QS-21 (N=6) | ACC-001 10 Micrograms (N=6) | ACC-001 10 Micrograms + QS-21 (N=6) | ACC-001 30 Micrograms (N=6) | ACC-001 30 Micrograms + QS-21 (N=6) | QS-21 (N=6) | Phosphate Buffered Saline (PBS) (N=4)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | ACC-001 3 Micrograms +QS-21 (N=6) | ACC-001 10 Micrograms (N=6) | ACC-001 10 Micrograms + QS-21 (N=6) | ACC-001 30 Micrograms (N=6) | ACC-001 30 Micrograms + QS-21 (N=6) | QS-21 (N=6) | Phosphate Buffered Saline (PBS) (N=4)
Cataract (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eyelid ptosis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 1
Duodenal polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tongue haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 2 | 3 | 2 | 1 | 2
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eosinophil count increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Glucose urine present (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prostatic specific antigen increased (Investigations) | 0/5 | 0/2 | 1/1 | 0/2 | 0/4 | 0/2 | 0/1
Protein urine present (Investigations) | 1 | 0 | 1 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mental impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abnormal sleep-related event (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abulia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aggression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Disinhibition (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paranoia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nephrocalcinosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aortic calcification (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.